CLINICAL TRIAL: NCT01199367
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of KW-2450 in Combination With Lapatinib and Letrozole in Subjects With Advanced or Metastatic Breast Cancer Whose Tumors Overexpress HER2
Brief Title: Safety, Tolerability, and Efficacy Study in Subjects With Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The results of the dose escalation phase did not identify a well-tolerated dose that would permit further study in Phase 2.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2450-US-002
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: advanced or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — KW-2450; Lapatinib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escallation (Experimental)
  Interventions: Drug: KW-2450 in combination with lapatinib and letrozole

INTERVENTIONS:
Drug: KW-2450 in combination with lapatinib and letrozole — Three subjects will be assigned to each of 4 sequential cohorts. Dose escalation may proceed once at least 3 subjects have completed 30 days of study treatment. Subjects who withdraw prior to completing Day 30 for reasons other than DLT will be replaced. If a DLT is observed, additional subjects may be enrolled so that up to 6 subjects are enrolled at that dose level.
  Other Names: KW-2450 lapatinib and letrozole

SUMMARY:
This study will determine the highest dose of KW-2450 in combination with lapatinib and letrozole that can be administered safely to subjects with advanced or metastatic breast cancer and to evaluate its effectiveness.

This study was terminated in Phase 1 and never proceeded to the Phase 2 portion of the study.

DETAILED DESCRIPTION:
This open-label, sequential, ascending, multi-dose, Phase 1/2 study will enroll up to 198 post-menopausal subjects with advanced or metastatic breast cancer whose tumors overexpress HER2. Subjects at each dose level will receive KW-2450 orally, on a continuous daily schedule in combination with lapatinib and letrozole.

In the Phase 1 portion of the study, dose escalation may proceed once ≥ 3 subjects have completed Day 30. The safety of each dose level will be established prior to enrollment of subjects in the next dose level. Dose escalation will proceed sequentially. Up to 6 subjects may be enrolled at each dose level. Enrollment will proceed until the MTD has been established or the highest dose level has been reached.

The Phase 2 portion of the trial will enroll 168 additional subjects. The dose level will be based on overall safety and tolerability assessments from the Phase 1 portion of the study. The subjects will be randomized into two treatment arms (1) Arm A, KW-2450 plus lapatinib plus letrozole: (2) Arm B, lapatinib plus letrozole.

This study was terminated in Phase 1 and never proceeded to the Phase 2 portion of the study.

ELIGIBILITY:
Inclusion Criteria

1. Histopathologically or cytologically confirmed, advanced or metastatic breast cancer (stage IIIb, IIIc or IV disease) including inflammatory breast cancer or inoperable locally advanced disease.
2. Documented ErbB2 overexpression
3. Estrogen receptor positive (ER+) and/or progesterone positive (PgR+) tumors
4. Measurable or non-measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria
5. A life expectancy of > 3 months for Phase 1 and > 6 months for Phase 2
6. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2 at study entry in Phase 1 and ≤ 1 in Phase 2;
7. Normal cardiac ejection fraction
8. Adequate hematologic, hepatic and renal function
9. Post-menopausal female (defined as the absence of a menstrual cycle for at least 12 consecutive months) or male subjects ≥ 18 years of age.
10. Sign an IRB or EC approved informed consent

Exclusion Criteria

1. Type 1 diabetes or uncontrolled Type 2 diabetes
2. Subjects showing clinical evidence or with a history of cataract(s), proliferate retinopathy or significant macular edema
3. Subjects with abnormal free T4 values and a history or evidence of thyroid disease
4. Subjects who are unable or unwilling to take metformin
5. Uncontrolled intercurrent illness
6. Known or suspected human immunodeficiency virus (HIV) infection or hepatitis B or C
7. Subjects with inflammatory diseases of the gastrointestinal tract
8. History of other malignancy. Subjects who have been disease free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible;
9. Subjects with extensive symptomatic visceral disease including hepatic involvement and pulmonary lymphangitic spread of tumor
10. A history of prior treatment with other agents specifically targeting IGFRs
11. Subjects who require pharmacological doses of glucocorticoids beyond replacement doses. The use of topical, intra-ocular or inhalation glucocorticoids is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To establish the safety, tolerability, and recommended Phase 2 dose of KW-2450 administered in combination with lapatinib and letrozole in subjects with previously treated or untreated advanced breast cancer. | 30 Days

SECONDARY OUTCOMES:
To determine the PK profile of KW-2450, lapatinib, and letrozole when administered together | 1 year (or until PD)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (5):
- United States (5):
  - Breastlink Research Group, Long Beach, California
  - Associates in Hematology-Oncology, Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - Clinical Oncology Associates, Farmington Hills, Michigan
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Dickson MA, P. LoRusso P, E. A. Sausville EA, Rao N, Kobayashi E, Kurman MR, Akinaga S, Schwartz GK. Open-label, sequential, ascending, multi-dose, phase I study of KW-2450 as monotherapy in subjects with previously treated advanced solid tumors. J Clin Oncol 29: 2011 (suppl; abstr 3078)